CLINICAL TRIAL: NCT07273331
Title: Quality of Life, Knowledge and Nursing Needs of Outpatients With Cirrhosis at Landspitali.
Brief Title: Nursing Needs of Patients With Cirrhosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Landspitali University Hospital (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Principal Investigator, Thora Jenny Gunnarsdottir, Professor, University of Iceland
Other Study IDs: LSH-44-2025
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Cirrhoses, Liver
Keywords: cross-sectional study,; nursing
MeSH Terms: interventions — Blood Specimen Collection; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — hemoglobin, platelets, white blood cell, ALP, AST, ALT, GGT, Bilirubin, Creatinine, Albumin, INR, Sodium, potassium, iron, iron binding capacity, ferritin, vitamin D, B-peth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with cirrhosis: patients with cirrhosis in outpatient clinic
  Interventions: Other: blood sample; Diagnostic Test: blood samples for analysis of cirrhosis

INTERVENTIONS:
Other: blood sample — measurement of blood status related to cirrhosis
  Other Names: interview
Diagnostic Test: blood samples for analysis of cirrhosis — interviews and blood sample taken

SUMMARY:
The primary objective of this study is to examine the quality of life, disease-related knowledge, and perceived nursing needs of adult patients diagnosed with liver cirrhosis who attend the outpatient clinic at Landspítali University Hospital. The study aims to generate clinically relevant insights that may inform improvements in nursing care and patient support. The research questions are: 1. what is the quality of life of patients with cirrhosis. 2. How do patients with cirrhosis describe their knowledge about the disease; and 3. How do patients with cirrhosis describe their nursing needs. Three questionnaires will be given to the patients. To assess quality of life Chronic Liver Disease Questionnaire (CLDQ) will be used. To validate knowledge and nursing needs two questionnaires will be used. The disease severity will be evaluated through clinical indicators such as MELD and Child-Pugh scores. In addition, the study will analyze demographic variables, including age, gender, education level, and employment status, to identify potential associations with quality of life, disease burden, and perceived care needs. By integrating clinical data, patient-reported outcomes, and sociodemographic factors, the study aims to support the development of evidence-based, individualized nursing strategies that enhance symptom management, reduce hospital admissions, and improve overall well-being for individuals living with liver cirrhosis in Iceland. The study has scientific value at national and international level, as it is based on a recognized measurement tool (CLDQ) and is in line with international emphasis on individualized treatment and early intervention in liver diseases. The results will provide deeper understanding of the quality of life and nursing needs of individuals with cirrhosis and support the development of targeted nursing services. The study can also shed light on the relationship between demographic factors and disease severity with service needs, as well as support policy development, education and improvements in the care of patients with chronic liver diseases. This study will have practical benefits for both patients and the Icelandic healthcare system. By identifying the specific nursing needs of individuals with cirrhosis, the study will support the development of targeted, individualized care plans that address symptom burden, disease progression, and psychosocial challenges. Improved nursing services, such as nutritional counseling, symptom management, and education about self-care of the disease, can improve patients' quality of life and promote greater independence.

DETAILED DESCRIPTION:
Cirrhosis is the end-stage of various liver diseases and has become increasingly prevalent in Europe due to rising obesity, excessive alcohol consumption, and undiagnosed liver diseases among marginalized groups, including immigrants (Karlsen et al., 2022). The EASL-Lancet Liver Commission report emphasizes that liver diseases are not only a medical issue but also a social and public health concern, reflecting and exacerbating inequalities in European healthcare systems (Karlsen et al., 2022). The report highlights that liver diseases are the second most common cause of working years lost in Europe, second only to ischemic heart disease, and that most deaths from liver diseases occur in working-age individuals. Despite many liver diseases being both preventable and treatable, diagnosis is often delayed, and treatment is provided at later stages, reducing quality of life and increasing healthcare costs. The EASL-Lancet report calls for a radical shift in the approach to liver health, emphasizing early diagnosis, prevention, and personalized care. Special emphasis is placed on the importance of nurses and other healthcare professionals in multidisciplinary teamwork, where nurses play a key role in education, support, and coordination of care. A nationwide population-based prospective study of cirrhosis in Iceland further supports these findings, revealing that the incidence of cirrhosis in Iceland has increased considerably during the last 4 decades and is currently comparable to other Western countries (Olafsson et al., 2021). Alcohol is still the leading cause, followed by metabolic-dysfunction associated steatotic liver disease (MASLD) and these two condition represent approximately two thirds of all etiologies in Iceland (Haraldsson et al. 2024). These studies underscores the need for effective management strategies and the critical role of healthcare professionals in improving patient outcomes. These insights particularly underscore the importance of developing nursing models in outpatient clinics that address the needs of patients with cirrhosis, focusing on quality of life, early intervention, and continuity of care. Many patients struggle with symptoms that disrupt daily activities and reduce independence, while uncertainty about disease progression adds to anxiety and feelings of vulnerability (Hansen et al., 2021). Nursing interventions have been shown to make a meaningful difference in the lives of patients with cirrhosis. Structured programs that focus on symptom monitoring, individualized education, and psychosocial support have improved patients´ experience of care and fostered a sense of empowerment (Hjorth et al., 2023). Nurse-led services are associated with fewer hospital readmissions and better long-term outcomes, as nurses are often able to detect subtle changes in patients´ conditions and intervene early to prevent complications (Kalo et al., 2023; Hjorth et al., 2025). In addition to clinical care, nurses provide vital emotional support, education, and advocacy, all of which are essential for maintaining an enhanced QoL.

The research plan, The study's design is cross-sectional in design and aims to recruit approximately 100-150 adult participants over a period of 10 months. Inclusion criteria are that participants must be 18 years of age or older with a confirmed diagnosis of cirrhosis, fluent in Icelandic or English. Exclusion criteria are severe cognitive impairment and serious or acute illness to ensure the reliability of self-reported data. Upon enrollment, participants will undergo a structured background interview to collect demographic data (age, gender, education level, employment status), disease perception, and symptom burden. This study utilizes three structured questionnaires to assess patient-reported outcomes related to quality of life, disease knowledge, and perceived nursing needs. The primary instrument is the Chronic Liver Disease Questionnaire (CLDQ), a validated tool specifically designed to evaluate quality of life in individuals with chronic liver conditions. The CLDQ covers six key domains: fatigue, emotional function, daily activity, abdominal symptoms, systemic symptoms, and worry related to illness. Each domain is assessed through multiple items that reflect the patient's experience over recent weeks. The questionnaire has demonstrated strong psychometric properties, including high internal consistency (Cronbach's alpha > 0.80), and has been approved for use in both Icelandic and English by the original author and publisher. In addition to the CLDQ, two custom-designed questionnaires were developed to address gaps in existing tools and to reflect the specific needs of patients with cirrhosis in the Icelandic healthcare context. The first, titled "Nursing Needs of Individuals with Liver Cirrhosis," consists of eleven statements addressing various aspects of nursing care and support. Participants indicate their level of agreement with each statement, which covers topics such as dietary guidance, symptom management, medication adherence, monitoring of weight and fluid retention, sleep and physical activity advice, emotional and social support, and access to nursing consultation. This instrument provides insight into patients' expectations and perceived gaps in outpatient nursing services. The second custom tool, "Knowledge of Liver Cirrhosis," is designed to assess patients' understanding of their condition. It includes eleven statements related to the causes, symptoms, diagnosis, treatment, and complications of cirrhosis, as well as the role of the liver in overall health. For each item, participants indicate whether the statement is true, false, or if they are unsure. Responses are scored to reflect the level of knowledge: no knowledge (0 points), low (1-3), moderate (4-6), good (7-9), and very good (10-11). This questionnaire aims to identify educational needs and inform targeted patient education strategies.

Clinical data, including diagnosis, complications, treatment history, and laboratory results, will be extracted from electronic health records. Participants will provide a blood sample during their outpatient visit. The sample will be used to assess liver function (ALP, ASAT, ALAT, GGT, bilirubin, albumin, INR), renal function (creatinine, sodium, potassium), hematological parameters (hemoglobin, white blood cells, platelets), iron status (iron, transferrin saturation), vitamin D levels, and B-Peth (phosphatidylethanol) as a biomarker of recent alcohol consumption. These results will be used to calculate MELD and Child-Pugh scores and to contextualize patient-reported outcomes. Blood sampling will be performed by trained clinical staff in accordance with standard hospital procedures. Data collection takes place during a planned outpatient visit. It begins with an interview according to an interview framework and an assessment of hepatic encephalopathy using animal testing. Disease severity will be calculated using MELD and Child-Pugh scores, based on both interview data and laboratory findings. Work and timeline: The study will start in November 2025 and end will be conducted for 20 months. Workpackage 1: Data collection will be done at Internal disease outpatient department in Landspitali where patients will come to participate from November 2025 - August 2026. Workpackage 2: will be analysis of data done with assistance from statistician from April 2026 to December 2026. Workpackage 3: July 2026 to June 2027 will be writing the final thesis done by master student. Workpackage 4: June 2027 to October 2027, writing manuscript for publication. The study has scientific value at the national and international level, as it is based on a recognized measurement tool (CLDQ) and is in line with international priorities for individualized treatment and early intervention in liver diseases. The results provide a deeper understanding of the quality of life and nursing needs of individuals with cirrhosis and support the development of targeted nursing services. The study will shed light on the relationship between demographic factors and disease severity with service needs, as well as support policy development, education and improvements in the care of patients with chronic liver diseases.

Management and co-operation This research is a collaboration between Landpitali University Hospital and University of Iceland, Faculty of Nursing and Midwifery and Faculty of Medicine. The study is managed by Dr. Þórunn Scheving Elíasdóttir, Associate Professor and Academic Chair of Anesthesia- and Perioperative Nursing at the University of Iceland, Faculty of Nursing and Midwifery.

Data management and publication of results in open access The results of the study will be used to support the development of outpatient nursing services for individuals with cirrhosis and to promote more targeted and individualized treatment. They will be published in a master's thesis at the University of Iceland and the aim is to publish them in both Icelandic and international open-access peer-reviewed journals in the field of nursing and health sciences. The results will also be presented at conferences related to health science research, both domestically and internationally, where the emphasis will be on communicating knowledge to professionals and supporting the clinical development of services for this patient group. The results will be published regardless of the outcome, in accordance with the ethics committee's rules of conduct.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for enrolment must meet the following criteria:

  * Be 18 years of age or older
  * Have a confirmed diagnosis of liver cirrhosis
  * Be fluent in Icelandic or English, to ensure participants can comprehend study materials and provide informed consent.

These criteria are designed to ensure that participants can meaningfully engage with the study procedures and provide reliable patient-reported data.

Exclusion Criteria:Participants will be excluded from the study if they meet any of the following conditions:

* Exhibit severe cognitive impairment that may interfere with informed consent or the completion of questionnaires
* Are experiencing acute or severe illness at the time of recruitment, such as recent hospitalization due to hepatic encephalopathy or bleeding from esophageal varices These exclusion criteria are intended to protect vulnerable individuals and maintain the integrity of the data collected.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cirrhosis in outpatient clinic at Landspitali
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Liver Disease Questionnaire score | November 2025 to End of August 2026
  score will be collected

CONTACTS AND LOCATIONS:
Locations (2):
- Iceland (2):
  - Eirberg Eiríksgata 34, Reykjavik
  - Faculty of Nursing and Midwifery, Reykjavik

IPD SHARING:
Plan to Share IPD: No
Will not be shared outside the researchers group in the study